CLINICAL TRIAL: NCT04374513
Title: SURVEY of RETAIL PHARMACISTS KNOWLEDGE, ROLE & BEHAVIOR DURING COVID-19 VIRUS OUTBREAK
Brief Title: Community Pharmacists Behaviour During Covid-19
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmacists and covid-19
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-04

CONDITIONS: Covid19
Keywords: Pharmacists/ covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the COVID-19 pandemic, governments issued movement restrictions and placed areas into quarantine to reduce the spread of the disease.Community pharmacists and their teams are a vital healthcare provider during the outbreak; they remain on the frontline of public health by serving as direct points of access for their patients. The retail pharmacists should provide public community, costumers and patients with right and trusted information about covid-19. They also should have role in awareness spreading regarding personnel safety and hygiene

DETAILED DESCRIPTION:
The survey will enroll as many community pharmacists as possible in the survey portion of the study - The number of participates have no limitations, at least 50 participants.

The survey will be enrolled in online google form, face to face interview & semi-structured telephone interviews if possible.

The research procedures:

1. An online survey link will include questions regarding the impact of role and behavior of retail pharmacists during covid-19 outbreak.
2. Face to face and semi-structured interviews if possible: For those pharmacists who state that they would like to participate in an interview, a random sample will be contacted.

Inclusion Criteria:

1. Post graduated pharmacist.
2. Community pharmacists.

Exclusion Criteria:

1. under graduated students.
2. not pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Post graduated pharmacist. Community pharmacists.

Exclusion Criteria:

* under graduated students. not pharmacist.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: community pharmacists
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
community pharmacists facing covid-19 | 6 months
  Evaluate the knowledge, role & behavior of retail pharmacists in facing covid-19 virus through the survey

CONTACTS AND LOCATIONS:
Overall Officials: Asser Ghoneim, phD, Principal Investigator — Professor in Pharmacology, Faculty of pharmacy, Damanhour University
Locations (2):
- Egypt (2):
  - Damanhour university, Beheira, Damanhour
  - Damanhour universty, Alexandria

REFERENCES:
- [Background] Farooq A, Laato S, Islam AKMN. Impact of Online Information on Self-Isolation Intention During the COVID-19 Pandemic: Cross-Sectional Study. J Med Internet Res. 2020 May 6;22(5):e19128. doi: 10.2196/19128. PMID 32330115
- [Background] Bukhari N, Rasheed H, Nayyer B, Babar ZU. Pharmacists at the frontline beating the COVID-19 pandemic. J Pharm Policy Pract. 2020 Apr 20;13:8. doi: 10.1186/s40545-020-00210-w. eCollection 2020. PMID 32328285
- [Background] Rutter V, Chan AHY, Tuck C, Bader L, Babar ZU, Bates I. Weaving the health and pharmaceutical care agenda through the themes of the commonwealth heads of government meeting (CHOGM), London 2018. J Pharm Policy Pract. 2018 Apr 11;11:10. doi: 10.1186/s40545-018-0140-3. eCollection 2018. PMID 29651337